CLINICAL TRIAL: NCT02318563
Title: A Multicenter, Randomized, Double-blind, Placebo- Controlled, Interventional Study to Assess the Safety and Efficacy of Pharmaceutical Cannabidiol Oral Solution as an Adjunctive Therapy for Treatment of Subjects With Inadequately Controlled Dravet Syndrome
Brief Title: Cannabidiol Oral Solution as an Adjunctive Therapy for Treatment of Participants With Inadequately Controlled Dravet Syndrome
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor elected not to continue with study.
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INS011-14-025
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Dravet Syndrome
Keywords: Treatment-resistant seizures
MeSH Terms: conditions — Epilepsies, Myoclonic | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol Oral Solution (Experimental): Participants will receive cannabidiol oral solution at an appropriate dose (no higher than 40 mg/kg/day) determined by data from a previous trial. The total daily dose will be administered in twice daily doses, approximately 12 hours apart.
  Interventions: Drug: Cannabidiol Oral Solution
- Placebo Solution (Placebo Comparator): Participants will receive matching placebo solution administered twice daily, approximately 12 hours apart.
  Interventions: Drug: Placebo Solution

INTERVENTIONS:
Drug: Cannabidiol Oral Solution — An oral solution containing pharmaceutical grade cannabidiol (nonplant-based)
  Arms: Cannabidiol Oral Solution
Drug: Placebo Solution — A matching oral solution containing no cannabidiol
  Arms: Placebo Solution

SUMMARY:
This Phase 3 study will enroll participants diagnosed with Dravet Syndrome (DS) who are still experiencing at least one tonic-clonic, clonic, and/or focal seizures with motor components (FSMC) per week, despite ongoing treatment with up to three antiepileptic drugs (AEDs), and meet the other inclusion/exclusion criteria.

Following a 28-day baseline period, participants will begin an 84-day treatment period. Participants will be assigned to receive twice-daily doses of placebo or cannabidiol oral solution at the highest dose determined to be safe in a previous trial.

Following study completion, all participants will be invited to receive Cannabidiol Oral Solution in an open label extension study (under a separate protocol).

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception, including clinical diagnosis of refractory DS and onset of seizures according to protocol-specified criteria
* Is able to speak and understand the language in which the study is being conducted, is able to understand the procedures and study requirements and has voluntarily signed and dated an informed consent form approved by the Institutional Review Board before the conduct of any study procedure
* In the opinion of the Investigator, the subject and/or parent(s)/caregiver(s) are able to keep accurate seizure diaries and the participant is able to take study drug and comply with the protocol, including dosing, medications and diet

Exclusion Criteria:

* Medical history is outside protocol-specified parameters
* Clinically significant history of allergic reactions or significant sensitivities to cannabinoids or to any of the other ingredients in the study drug
* Inadequate supervision by parents or guardians
* History or current use of dietary supplements, drugs or over-the counter medications outside protocol-specified parameters
* Signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise: 1) the safety or well-being of the participant or study staff; 2) the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding); 3) the analysis of results

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-30 (Estimated); Primary Completion 2018-06-17 (Estimated); Study Completion 2018-06-17 (Estimated)

PRIMARY OUTCOMES:
Percent change in the frequency of tonic-clonic, clonic, and focal seizures with motor components | Data point for observation period to data point for treatment period Weeks 9 through 12

SECONDARY OUTCOMES:
Percent change from baseline in the severity of tonic-clonic, clonic, and focal seizures with motor components | Data point for observation period to data point for treatment period Weeks 9 through 12
Percent change from baseline in the duration of tonic-clonic, clonic, and focal seizures with motor components | Data point for observation period to data point for treatment period Weeks 9 through 12
Percent change from baseline in the frequency of all seizure activity independent of seizure type | Data point for observation period to data point for treatment period Weeks 9 through 12
Change from baseline in parent(s)/caregiver(s) Clinical Global Impressions of Improvement (CGI-I) | Data point for observation period to data point for treatment period Weeks 9 through 12
Change from baseline in parent(s)/caregiver(s) Clinical Global Impressions of Severity (CGI-S) | Data point for observation period to data point for treatment period Weeks 9 through 12
Change from baseline in Investigator CGI-I | Data point for observation period to data point for treatment period Weeks 9 through 12
Change from baseline in Investigator CGI-S | Data point for observation period to data point for treatment period Weeks 9 through 12

CONTACTS AND LOCATIONS:
Overall Officials: Neha Parikh, Study Director — INSYS Therapeutics Inc